CLINICAL TRIAL: NCT01172522
Title: A Pilot Randomized Double Blind Study to Assess the Safety and Efficacy of 1% Ibuprofen/ 1%Fexofenadine Topical Cream for the Treatment of Dark Circles Under the Eyes
Brief Title: Topical Treatment of Under Eye Dark Circles and Swelling
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Connecticut Sinus Center, PC (Other)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS910510
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Results first posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Edema
Keywords: Under eye dark circles; Under eye puffiness
MeSH Terms: conditions — Edema | interventions — fexofenadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fexofenadine left; placebo right (Experimental): Topical treatment active versus placebo.
  Double blind randomized placebo controlled split face intrasubject comparison.
  Interventions: Drug: Fexofenadine; Drug: Placebo
- Fexofenadine right; placebo left (Experimental): Split face double blind
  Interventions: Drug: Fexofenadine; Drug: Placebo

INTERVENTIONS:
Drug: Fexofenadine — Fexofenadine 1%
  Other Names: Topical fexofenadine
Drug: Placebo — Placebo
  Other Names: Topical placebo

SUMMARY:
This study examines topical treatment of under eye circles and swelling.

DETAILED DESCRIPTION:
This study examines topical treatment of under eyes dark circles and under eye swelling.

ELIGIBILITY:
Inclusion Criteria:

* Under eye dark circles and swelling

Exclusion Criteria:

* Under age 18
* Allergy to tested medicines

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward M Lane, MD, Study Director — The Connecticut Sinus Center, PC
Locations (1):
- TKL Research, Paramus, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fexofenadine Right Side; Placebo Left Side: Topical treatment active versus placebo.
  Double blind randomized placebo controlled split face intrasubject comparison. Participants were randomized to side of face with active drug versus side of face with control, but with each treatment going on concurrently.
- Fexofenadine Left Side; Placebo Right Side: Subjects were randomized as to side of face treated with test article versus placebo
Period: Overall Study
Arm/Group | Fexofenadine Right Side; Placebo Left Side | Fexofenadine Left Side; Placebo Right Side
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adult with evidence of dark peri-orbital areas
Groups:
- Fexofenadine Right Side; Placebo Left Side: Topical treatment active versus placebo.
  Double blind randomized placebo controlled split face intrasubject comparison.
  Placebo, fexofenadine
- Fexofenadine Left Side; Placebo Right Side: Topical treatment active versus placebo.
  Double blind randomized placebo controlled split face intrasubject comparison.
  Fexofenadine, placebo
- Total: Total of all reporting groups
Arm/Group | Fexofenadine Right Side; Placebo Left Side | Fexofenadine Left Side; Placebo Right Side | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (15) | 30 (15) | 30 (15)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Showed Improvement in Under Eye Swelling and Dark Circles Relative to Baseline Per Intervention
Description: Efficacy was measured per intervention by assessing number of participants with improvement in under eye dark circles and swelling. Criteria used to assess under eye improvement and swelling was by a 5 point scale comparing each week's photographic appearance to the appearance at baseline: 1) fexofenadine right and placebo left, and 2) fexofenadine left and placebo right. The split face comparison was noted in efficacy measured changes in under eye swelling and dark circles relative to baseline. Participants were graded by 2 blinded dermatologists who reviewed photographs of all participants at entry and weekly until end of study plus one week, day 37. Total number of participants: 30. Placebo right and fexofenadine left 15 participants. Placebo left and fexofenadine right 15 participants.
Time Frame: Baseline, weekly, and end of study +7 days
Population: Thirty participants in total; 15 had fexofenadine left and placebo right; 15 had fexofenadine right and placebo left.
Measure: Number; unit: participants
Groups:
- Fexofenadine: All participants that received fexofenadine
- Placebo: All participants that received placebo
Arm/Group | Fexofenadine | Placebo
Number analyzed (Participants) | 30 | 30
participants | 0 | 0
Statistical Analysis 1: Comparison: Fexofenadine vs Placebo; Test type: Superiority or Other; p = 1, Chi-squared; Other = 0 — P values above 0.05 is considered statistically insignificant in this study

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Split Face Intrasubject Comparison: Topical treatment active versus placebo
  Double blind randomized placebo controlled split face intrasubject comparison.
Arm/Group | Split Face Intrasubject Comparison
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes